CLINICAL TRIAL: NCT00552851
Title: Changes of Left Ventricular Mass and Cardiac Function in Patients With Active Acromegaly During Treatment With the Growth Hormone Receptor Antagonist Pegvisomant: an Open-labelled, Prospective Study
Brief Title: Changes of Left Ventricular Mass and Cardiac Function in Patients With Active Acromegaly During Treatment With the Growth Hormone Receptor Antagonist Pegvisomant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Prof. Bruno Allolio, Department of Endocrinology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRA 6290010; EudraCT No: 2006-001108-35
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Acromegaly; Heart Failure; Hypertrophy, Left Ventricular
Keywords: acromegaly; heart failure; hypertrophy; cardiomegaly
MeSH Terms: conditions — Acromegaly; Heart Failure; Hypertrophy, Left Ventricular; Hypertrophy; Cardiomegaly | interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pegvisomant (Other): patients with active acromegaly and impaired cardiac function
  Interventions: Drug: pegvisomant

INTERVENTIONS:
Drug: pegvisomant — booster dosage 80 mg once sc., than 10 mg once per day, uptitration in steps of 5 mg up to an IGF-1 level in the normal range (every 4 weeks), max. 30 mg once per day. Duration of treatment: one year
  Other Names: Somavert

SUMMARY:
The purpose of this study is to evaluate changes in left ventricular mass and cardiac function in patients with active acromegaly before and after treatment with the growth hormone receptor antagonist pegvisomant for one year.

ELIGIBILITY:
Inclusion Criteria:

* Active acromegaly in adult subjects (≥ 18 years) after surgery and/or radiation therapy with elevated IGF-1 levels despite treatment with somatostatin analogues or dopamine agonists
* Pegvisomant therapy is indicated (i. e. patients who have had an inadequate response to surgery and/or radiation therapy and/or other medical therapy, or for whom these therapies are not appropriate)
* Evidence of left ventricular hypertrophy (infero-lateral wall thickness ≥ 12 mm assessed by echocardiography) or
* Evidence of impaired diastolic function (≥ stage 2 as assessed by echocardiography) or
* Evidence of systolic dysfunction (Ejection fraction < 50% assessed by echocardiography)
* Stable medication for arterial hypertension and heart failure for 3 months
* Written informed consent.

Exclusion Criteria:

* Pregnancy and lactation period
* Previous therapy with Pegvisomant
* Suspected or known hypersensitivity to the drug or any of its components
* Contraindications for MRI
* History of malignancy during the last 5 years
* Suspected or known drug or alcohol abuse
* Patients who are neither able to self administer study medication on a daily basis nor have a caregiver who can administer study medication to the patient on a daily basis
* Any condition which in the opinion of the investigator makes the patient unsuitable for inclusion
* Participation in another clinical trial
* Pituitary adenoma with a distance to the optic chiasm of < 3 mm
* Any other drug for treatment of acromegaly (e.g. dopamine agonists, Somatostatin analogues) which would be necessary during the study or patients who apply for radiotherapy
* Instable heart insufficiency classified as NYHA IV.
* Severe renal insufficiency, liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2006-06; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Change in peak systolic strain rate (SRSYS) determined by Color Doppler Myocardial Imaging (CDMI). | one year

SECONDARY OUTCOMES:
Ejection fraction,Enddiastolic thickness of the infero-lateral wall,Diastolic function,Left ventricular mass index,Stroke volume,Ejection fraction (MRI),CO,Late hyperenhancement,IGF-I,insulin sensitivity,Ringsize,adverse events,Endothelial function | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Principal Investigator — University of Wuerzburg. Department of Endocrinology
Locations (1):
- University of Wuerzburg, Department of Endocrinology, Würzburg, Bavaria, Germany